CLINICAL TRIAL: NCT02983942
Title: Ketogenic Diet Adjunctive to High Dose Methotrexate Chemotherapy for Primary Central Nervous System Lymphoma
Brief Title: Ketogenic Diet Adjunctive to HD-MTX Chemotherapy for Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Song Lin, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0010
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: ketogenic diet; Primary Central Nervous System Lymphoma; chemotherapy
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketogenic diet group (Experimental): Ketogenic diet is given in combination to standard HD-MTX chemotherapy to primary central nervous system lymphoma patients. Blood ketone is kept no less than 2mmol/L during the initial 4 cycles of chemotherapy. The adverse events is monitored and recorded. Tumor response is evaluated and recorded.
  Interventions: Dietary Supplement: ketogenic diet
- routine diet group (Active Comparator): Standard HD-MTX chemotherapy is given with routine diet.Blood ketone is measured and recorded. The adverse events is monitored and recorded. Tumor response is evaluated and recorded.
  Interventions: Dietary Supplement: Routine diet

INTERVENTIONS:
Dietary Supplement: ketogenic diet — Ketogenic diet is given to maintain blood ketone level above 2 mmol/L.
  Arms: ketogenic diet group
Dietary Supplement: Routine diet — Routine diet is given without blood ketone requirement
  Arms: routine diet group

SUMMARY:
Ketogenic diet has shown auxiliary effect on treatment of malignant tumors require high glucose consumption. This study is designed to evaluate the safety and efficacy of ketogenic diet adjunctive to high dose methotrexate(HD-MTX) chemotherapy for primary central nervous system lymphoma (PCNSL).

DETAILED DESCRIPTION:
In a pilot study of primary central nervous system(CNS) lymphoma patients, ketogenic diet was given in adjunction with standard HD-MTX chemotherapy as interventional group; standard HD-MTX is given with routine diet as control group. The primary endpoint is the safety of ketogenic diet in PCNSL patients receiving chemotherapy, secondary endpoints include rate of complete remission, remission time, rate of tumor relapse and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Histopathologically confirmed PCNSL
3. No systemic involvement
4. Ability and willingness to sign informed consent
5. Normal liver and kidney function
6. Karnofsky Performance Score of 60 or more

Exclusion Criteria:

1. Any systemic involvement of the tumor
2. Systemic illness or medical condition may pose additional risk, including cardiac, metabolic or endocrine disorders; incompensated renal or liver disfunction; history of renal calculi, hyperuricemia, hyper calcemia, mitochondrial disease, known disorder of fatty acid metabolism, porphyria, carnitine deficiency and pancreatitis
3. Uncontrolled hyperlipidemia or hyperglycemia
4. Human immunodeficiency virus positive, or hepatitis C positive
5. Pregnancy of breastfeeding
6. Inability or unwillingness to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v4.0 | Two years
  The number and incidence (%) of treatment related adverse events among participants

SECONDARY OUTCOMES:
The chemosensitivity of tumor | Two years
  The rate of complete remission after treatment assessed according to serial contrast Magnetic Resonance Imaging (MRI)
Long term effect of chemotherapy | Two years
  The average time from complete remission of tumor to relapse
overall survival | Three years
  Participants will be followed until reported death to calculate overall survival
Quality of life | Two years
  Short Form 36 Questionnaire will be used to assess patients' quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Song Lin, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided